CLINICAL TRIAL: NCT04476004
Title: Effects of Electromyographic Visual Feedback for Spinal Accessory Nerve Dysfunction in Oral Cancer Survivors With Neck Dissection: a Randomized Clinical Trial
Brief Title: Effects of Electromyographic Visual Feedback for Spinal Accessory Nerve Dysfunction After Neck Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201901788A3
Record Dates: First submitted 2020-07-16; First posted 2020-07-17 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2020-10

CONDITIONS: Oral Cancer
Keywords: Scapular-focused exercise; Scapular Dyskinesis; Spinal accessory nerve; Physical therapy; Electromyography; Visual feedback
MeSH Terms: conditions — Mouth Neoplasms | interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): EMG group
  Interventions: Other: scapular-focused exercise; Other: visual feedback
- control group (Active Comparator): exercise group
  Interventions: Other: scapular-focused exercise

INTERVENTIONS:
Other: scapular-focused exercise — scapular-focused exercise
Other: visual feedback — EMG visual feedback
  Arms: experimental group

SUMMARY:
Patients with head and neck cancer and undergo neck dissection often suffer from spinal accessory nerve dysfunction (e.g. shoulder droop, shoulder pain, and decreased active range of motion (AROM) of the shoulder joint and scapular muscle strength), even the spinal accessory nerve is preserved during surgery. Abnormal muscle activities of scapular muscles, including upper trapezius (UT), middle trapezius (MT), lower trapezius (LT), serratus anterior (SA) and rhomboid were reported in subsequent research articles. Particularly for the trapezius muscle, the decreased amplitudes were observed even after 9 months of neck dissection. It has been reported that conscious correction of scapular orientation during arm movement could increase trapezius muscle activities, and motor control training could change scapular kinematic such as increased posterior tilt and upward rotation during arm movement.

DETAILED DESCRIPTION:
Patients with head and neck cancer and undergo neck dissection often suffer from spinal accessory nerve dysfunction (e.g. shoulder droop, shoulder pain, and decreased active range of motion (AROM) of the shoulder joint and scapular muscle strength), even the spinal accessory nerve is preserved during surgery. Abnormal muscle activities of scapular muscles, including upper trapezius (UT), middle trapezius (MT), lower trapezius (LT), serratus anterior (SA) and rhomboid were reported in subsequent research articles. Particularly for the trapezius muscle, the decreased amplitudes were observed even after 9 months of neck dissection. It has been reported that conscious correction of scapular orientation during arm movement could increase trapezius muscle activities, and motor control training could change scapular kinematic such as increased posterior tilt and upward rotation during arm movement.

The aim of this study is to explore the effects of electromyographic (EMG) visual feedback on scapular muscle activities and strength in oral cancer survivors with spinal accessory nerve dysfunction. Investigators will recruit 60 newly diagnosed oral cancer subjects through the plastic surgeon's referral from January 2020 to February 2021. The participants will be randomized separated into experimental or control group. Each group would receive regular physical therapy for shoulder function (e.g. transcutaneous electrical stimulation, shoulder joint range of motion exercise) and scapular-focused exercise. EMG visual feedback would be combined with scapular-focused exercise.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed oral cancer subjects with neck dissection
* age between 20 and 65 years
* having the clinical signs of neck-dissection related shoulder dysfunction (e.g. shoulder droop, limited AROM of shoulder abduction, and insufficient muscle strength of shoulder abduction to against gravity)

Exclusion Criteria:

* were pregnant or breastfeeding
* had distant metastasis or recurrence
* were unable to communicate or comprehend the questionnaires
* had a history of shoulder dysfunction before neck dissection (e.g. shoulder pain, tendinitis, tendon rupture, shoulder capsulitis, or neuropathy)
* had any disorder that could influence movement performance
* bilateral neck dissection

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
shoulder pain | 0, 3 months
  Visual Analog Scale, total range=0-10, 0 means no pain and 10 means the obvious pain
shoulder joint range of motion | 0, 3 months
  abduction measured by goniometer, total range: 0-180
scapular position | 0, 3 months
  Modified Lateral Scapular Slide Test

SECONDARY OUTCOMES:
quality of life C-30 | 0, 3 months
  European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30, total range= 0-100. A higher score on the functional scale or global health scale represents a higher level of functioning or quality of life.
shoulder function | 3 months
  The Disabilities of the Arm, Shoulder and Hand (DASH) Score, total range: 0-100. Higher scores indicate greater disability.
muscle activity to perform arm movement | 3 months
  EMG activities measure the muscle activities of the upper trapezius, middle trapezius, and lower trapezius
maximal isometric muscle strength (MVIC) | 3 months
  measurement of MVIC of the upper trapezius, middle trapezius, and lower trapezius
EMG activities of maximal isometric muscle strength (MVIC) | 3 months
  measurement of surface EMG activities of the upper trapezius, middle trapezius, and lower trapezius during MVIC

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, Master, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Plastic and Reconstructive Surgery Rehabilitation Center, Chung Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Result] Wong CH, Wei FC. Microsurgical free flap in head and neck reconstruction. Head Neck. 2010 Sep;32(9):1236-45. doi: 10.1002/hed.21284. PMID 20014446
- [Result] Lutz BS, Wei FC. Microsurgical workhorse flaps in head and neck reconstruction. Clin Plast Surg. 2005 Jul;32(3):421-30, vii. doi: 10.1016/j.cps.2005.02.006. PMID 15979480
- [Result] Sheikh A, Shallwani H, Ghaffar S. Postoperative shoulder function after different types of neck dissection in head and neck cancer. Ear Nose Throat J. 2014 Apr-May;93(4-5):E21-6. PMID 24817237
- [Result] van der Molen L, van Rossum MA, Burkhead LM, Smeele LE, Rasch CR, Hilgers FJ. A randomized preventive rehabilitation trial in advanced head and neck cancer patients treated with chemoradiotherapy: feasibility, compliance, and short-term effects. Dysphagia. 2011 Jun;26(2):155-70. doi: 10.1007/s00455-010-9288-y. Epub 2010 Jul 11. PMID 20623305
- [Result] Eades M, Murphy J, Carney S, Amdouni S, Lemoignan J, Jelowicki M, Nadler M, Chasen M, Gagnon B. Effect of an interdisciplinary rehabilitation program on quality of life in patients with head and neck cancer: review of clinical experience. Head Neck. 2013 Mar;35(3):343-9. doi: 10.1002/hed.22972. Epub 2012 Mar 16. PMID 22422558
- [Result] McGarvey AC, Osmotherly PG, Hoffman GR, Chiarelli PE. Impact of neck dissection on scapular muscle function: a case-controlled electromyographic study. Arch Phys Med Rehabil. 2013 Jan;94(1):113-9. doi: 10.1016/j.apmr.2012.07.017. Epub 2012 Aug 1. PMID 22864015
- [Result] Stubblefield MD. Radiation fibrosis syndrome: neuromuscular and musculoskeletal complications in cancer survivors. PM R. 2011 Nov;3(11):1041-54. doi: 10.1016/j.pmrj.2011.08.535. PMID 22108231
- [Result] Chan JY, Lua LL, Starmer HH, Sun DQ, Rosenblatt ES, Gourin CG. The relationship between depressive symptoms and initial quality of life and function in head and neck cancer. Laryngoscope. 2011 Jun;121(6):1212-8. doi: 10.1002/lary.21788. Epub 2011 May 3. PMID 21541945
- [Result] EWING MR, MARTIN H. Disability following radical neck dissection; an assessment based on the postoperative evaluation of 100 patients. Cancer. 1952 Sep;5(5):873-83. doi: 10.1002/1097-0142(195209)5:53.0.co;2-4. No abstract available. PMID 12988177
- [Result] McNeely ML, Parliament MB, Seikaly H, Jha N, Magee DJ, Haykowsky MJ, Courneya KS. Effect of exercise on upper extremity pain and dysfunction in head and neck cancer survivors: a randomized controlled trial. Cancer. 2008 Jul 1;113(1):214-22. doi: 10.1002/cncr.23536. PMID 18457329
- [Result] McNeely ML, Parliament M, Courneya KS, Seikaly H, Jha N, Scrimger R, Hanson J. A pilot study of a randomized controlled trial to evaluate the effects of progressive resistance exercise training on shoulder dysfunction caused by spinal accessory neurapraxia/neurectomy in head and neck cancer survivors. Head Neck. 2004 Jun;26(6):518-30. doi: 10.1002/hed.20010. PMID 15162353
- [Result] Carr SD, Bowyer D, Cox G. Upper limb dysfunction following selective neck dissection: a retrospective questionnaire study. Head Neck. 2009 Jun;31(6):789-92. doi: 10.1002/hed.21018. PMID 19260131
- [Result] Dijkstra PU, van Wilgen PC, Buijs RP, Brendeke W, de Goede CJ, Kerst A, Koolstra M, Marinus J, Schoppink EM, Stuiver MM, van de Velde CF, Roodenburg JL. Incidence of shoulder pain after neck dissection: a clinical explorative study for risk factors. Head Neck. 2001 Nov;23(11):947-53. doi: 10.1002/hed.1137. PMID 11754498
- [Result] Erisen L, Basel B, Irdesel J, Zarifoglu M, Coskun H, Basut O, Tezel I, Hizalan I, Onart S. Shoulder function after accessory nerve-sparing neck dissections. Head Neck. 2004 Nov;26(11):967-71. doi: 10.1002/hed.20095. PMID 15459926
- [Result] Lima LP, Amar A, Lehn CN. Spinal accessory nerve neuropathy following neck dissection. Braz J Otorhinolaryngol. 2011 Mar-Apr;77(2):259-62. doi: 10.1590/s1808-86942011000200017. PMID 21537629
- [Result] Umeda M, Shigeta T, Takahashi H, Oguni A, Kataoka T, Minamikawa T, Shibuya Y, Komori T. Shoulder mobility after spinal accessory nerve-sparing modified radical neck dissection in oral cancer patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jun;109(6):820-4. doi: 10.1016/j.tripleo.2009.11.027. Epub 2010 Mar 17. PMID 20299249
- [Result] Worsley P, Warner M, Mottram S, Gadola S, Veeger HE, Hermens H, Morrissey D, Little P, Cooper C, Carr A, Stokes M. Motor control retraining exercises for shoulder impingement: effects on function, muscle activation, and biomechanics in young adults. J Shoulder Elbow Surg. 2013 Apr;22(4):e11-9. doi: 10.1016/j.jse.2012.06.010. Epub 2012 Sep 1. PMID 22947240
- [Result] Huang TS, Du WY, Wang TG, Tsai YS, Yang JL, Huang CY, Lin JJ. Progressive conscious control of scapular orientation with video feedback has improvement in muscle balance ratio in patients with scapular dyskinesis: a randomized controlled trial. J Shoulder Elbow Surg. 2018 Aug;27(8):1407-1414. doi: 10.1016/j.jse.2018.04.006. Epub 2018 Jun 6. PMID 29886062
- [Result] Roy JS, Moffet H, Hebert LJ, Lirette R. Effect of motor control and strengthening exercises on shoulder function in persons with impingement syndrome: a single-subject study design. Man Ther. 2009 Apr;14(2):180-8. doi: 10.1016/j.math.2008.01.010. Epub 2008 Mar 20. PMID 18358760
- [Result] Shepherd KL, Fisher SE. Prospective evaluation of quality of life in patients with oral and oropharyngeal cancer: from diagnosis to three months post-treatment. Oral Oncol. 2004 Aug;40(7):751-7. doi: 10.1016/j.oraloncology.2004.01.018. PMID 15172646
- [Result] Schliephake H, Jamil MU. Prospective evaluation of quality of life after oncologic surgery for oral cancer. Int J Oral Maxillofac Surg. 2002 Aug;31(4):427-33. doi: 10.1054/ijom.2001.0194. PMID 12361079
- [Result] Barrios R, Bravo M, Gil-Montoya JA, Martinez-Lara I, Garcia-Medina B, Tsakos G. Oral and general health-related quality of life in patients treated for oral cancer compared to control group. Health Qual Life Outcomes. 2015 Jan 23;13:9. doi: 10.1186/s12955-014-0201-5. PMID 25613348
- [Result] McNeely ML, Parliament MB, Seikaly H, Jha N, Magee DJ, Haykowsky MJ, Courneya KS. Sustainability of outcomes after a randomized crossover trial of resistance exercise for shoulder dysfunction in survivors of head and neck cancer. Physiother Can. 2015 Winter;67(1):85-93. doi: 10.3138/ptc.2014-13O. PMID 25931658
- [Result] Ch'ng S, Oates J, Gao K, Foo K, Davies S, Brunner M, Clark JR. Prospective quality of life assessment between treatment groups for oral cavity squamous cell carcinoma. Head Neck. 2014 Jun;36(6):834-40. doi: 10.1002/hed.23387. Epub 2013 Sep 2. PMID 23720248
- [Result] Curtis T, Roush JR. The Lateral Scapular Slide Test: A Reliability Study of Males with and without Shoulder Pathology. N Am J Sports Phys Ther. 2006 Aug;1(3):140-6. PMID 21522226
- [Result] McGarvey AC, Osmotherly PG, Hoffman GR, Chiarelli PE. Scapular muscle exercises following neck dissection surgery for head and neck cancer: a comparative electromyographic study. Phys Ther. 2013 Jun;93(6):786-97. doi: 10.2522/ptj.20120385. Epub 2013 Feb 21. PMID 23431215
- [Result] Kibler WB, Ludewig PM, McClure PW, Michener LA, Bak K, Sciascia AD. Clinical implications of scapular dyskinesis in shoulder injury: the 2013 consensus statement from the 'Scapular Summit'. Br J Sports Med. 2013 Sep;47(14):877-85. doi: 10.1136/bjsports-2013-092425. Epub 2013 Apr 11. PMID 23580420
- [Result] Baskurt Z, Baskurt F, Gelecek N, Ozkan MH. The effectiveness of scapular stabilization exercise in the patients with subacromial impingement syndrome. J Back Musculoskelet Rehabil. 2011;24(3):173-9. doi: 10.3233/BMR-2011-0291. PMID 21849731
- [Result] Struyf F, Nijs J, Mollekens S, Jeurissen I, Truijen S, Mottram S, Meeusen R. Scapular-focused treatment in patients with shoulder impingement syndrome: a randomized clinical trial. Clin Rheumatol. 2013 Jan;32(1):73-85. doi: 10.1007/s10067-012-2093-2. Epub 2012 Oct 2. PMID 23053685
- [Result] Park SI, Choi YK, Lee JH, Kim YM. Effects of shoulder stabilization exercise on pain and functional recovery of shoulder impingement syndrome patients. J Phys Ther Sci. 2013 Nov;25(11):1359-62. doi: 10.1589/jpts.25.1359. Epub 2013 Dec 11. PMID 24396188
- [Result] Moezy A, Sepehrifar S, Solaymani Dodaran M. The effects of scapular stabilization based exercise therapy on pain, posture, flexibility and shoulder mobility in patients with shoulder impingement syndrome: a controlled randomized clinical trial. Med J Islam Repub Iran. 2014 Aug 27;28:87. eCollection 2014. PMID 25664288
- [Result] Turgut E, Duzgun I, Baltaci G. Effects of Scapular Stabilization Exercise Training on Scapular Kinematics, Disability, and Pain in Subacromial Impingement: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Oct;98(10):1915-1923.e3. doi: 10.1016/j.apmr.2017.05.023. Epub 2017 Jun 24. PMID 28652066
- [Result] Nowotny J, Kasten P, Kopkow C, Biewener A, Mauch F. Evaluation of a New Exercise Program in the Treatment of Scapular Dyskinesis. Int J Sports Med. 2018 Oct;39(10):782-790. doi: 10.1055/a-0608-4584. Epub 2018 Aug 27. PMID 30149414
- [Result] De Mey K, Danneels LA, Cagnie B, Huyghe L, Seyns E, Cools AM. Conscious correction of scapular orientation in overhead athletes performing selected shoulder rehabilitation exercises: the effect on trapezius muscle activation measured by surface electromyography. J Orthop Sports Phys Ther. 2013 Jan;43(1):3-10. doi: 10.2519/jospt.2013.4283. Epub 2012 Nov 16. PMID 23160271
- [Derived] Chen YH, Liang WA, Lin CR, Huang CY. A randomized controlled trial of scapular exercises with electromyography biofeedback in oral cancer patients with accessory nerve dysfunction. Support Care Cancer. 2022 Oct;30(10):8241-8250. doi: 10.1007/s00520-022-07263-4. Epub 2022 Jul 11. PMID 35821447